CLINICAL TRIAL: NCT03860233
Title: Benefits of Oxytocin in OSA Patients Using CPAP
Brief Title: Benefits of Oxytocin in Obstructive Sleep Apnea (OSA) Patients Using Continuous Positive Airway Pressure (CPAP) Machine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vivek Jain (Other)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor-Investigator, Vivek Jain, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GWU_IRB_031857
Record Dates: First submitted 2019-01-24; First posted 2019-03-01 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive
Keywords: Continuous Positive Airway Pressure; CPAP; Oxytocin
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All study staff are masked except the pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visit 1 Randomization (Experimental): At visit 1subjects will receive one of two interventions: either Oxytocin Intranasal spray (40 IU) or Placebo Intranasal spray. Subjects will be blinded as to which drug they are receiving.
  Interventions: Drug: Oxytocin; Drug: Placebo
- Visit 2 Crossover Randomization (Experimental): At visit 2 subjects will receive the opposite intervention from the one they received at visit 1: either Oxytocin Intranasal spray (40 IU) or Placebo Intranasal spray. Subjects will be blinded as to which drug they are receiving.
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 40 IU administered intranasal, within 1 hour prior to sleeping for 14 days
Drug: Placebo — Intranasal spray to mimic Oxytocin intranasal spray
  Other Names: Placebo (for Oxytocin)

SUMMARY:
This study will investigate if an intra-nasal nose spray of the drug oxytocin can decrease the amount of pressure needed from the automatic Continuous Positive Airway Pressure (CPAP) device while sleeping decreasing some of the harmful effects of low oxygen in people with sleep apnea.

This study will last 35 nights and involves spending three nights in the sleep lab at George Washington University. There are no additional costs to participants and no compensation for being involved in the study.

DETAILED DESCRIPTION:
This is a rigorous randomized, double-blinded, cross-over study. Patients will self-administer either oxytocin nasal spray (40IU/ml), or sterile water spray, for 2 weeks, followed by 2 weeks of the spray not used initially (with a one week washout period in between). Subjects will have been using (for a minimum of 1 month) an auto-adjusting/titrating positive airway pressure (auto-CPAP device) as this is the mainstay of treatment for OSA and considered standard-of-care. All auto-CPAP devices are capable of recording frequency and duration of patient use (thus helping with compliance monitoring) and also recording the pressure needed to keep the airway open.

After obtaining consent, forty subjects will undergo the following (at Day 1): (a) venipuncture to obtain 50 ml of blood (to be stored for use to analyze inflammatory markers and biomarkers of oxidative stress, (b) an overnight sleep study in the sleep-lab (with their auto-CPAP) to assess sleep architecture, (c) download of their compliance report from the auto-CPAP to assess mean PAP pressure. They will then be randomized to receive either 40 i.u (1 ml/10 nasal sprays) intranasally of oxytocin per night for 2 weeks (14 days), or matching placebo (1 ml/10 sprays) intranasally per night for 2 weeks (14 days). The researchers and subjects will be blinded to the order of oxytocin versus placebo and to the randomization process (will be done by the MFA-investigational drug pharmacy). The end of the 2 week (14 day) period will mark day 14. Subjects will continue using their auto-CPAP during these 2 weeks as per standard-of-care. At day 14: (a) subjects will undergo another overnight in-lab sleep study (with their auto-CPAP) to assess sleep architecture, and (b) have another venipuncture to collect 50 ml of blood, (c) download of compliance report from their auto-CPAP, and continue to take either the placebo or oxytocin. Each subject will then have a wash-out period of 1 week (Days 14-21, they will continue using their auto-CPAP during this week as per standard-of-care). Beginning at Day 21 each subject will then receive either oxytocin or placebo (the opposite of what they did not receive the first time at point A) for 14 days (2 weeks) Days 21-35: nightly dose of either 40 i.u of oxytocin (1 ml/10 sprays) or matching placebo intranasally after a wash out period of 1 week (days 14-21). Again, the researchers and subjects will be blinded to the compound given to the subjects. Subjects will continue using their auto-CPAP during these 2 weeks as per standard-of-care. At the end of this 2 week period will be day 35, when subjects will undergo another overnight in-lab sleep study and continue to take either the placebo or oxytocin (with their auto-CPAP) to assess sleep architecture, have another venipuncture to collect 50 ml of blood, and we will download the compliance report and pressure data from their auto-CPAP. The subject and all investigators will be blinded to the sequence of oxytocin or placebo until the study is unblinded at the end of the 35 day protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age or older.

Exclusion Criteria:

* subjects not willing to or otherwise unable to use CPAP for treatment of OSA.
* Presence of other sleep disorders
* Pregnant or breastfeeding women
* Women of child-bearing age (WOCBA) not willing or unable to use an accepted method to avoid pregnancy for the entire duration of the study
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detain or treatment of either a psychiatric or physical (i.e. infectious disease) illness
* Patients unable to give consent because of a language barrier, or other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Use of oxytocin will change pressure required to keep open airway during auto-CPAP use | 5 weeks
  CPAP pressures will be monitored during study via electronic data retrieval system

SECONDARY OUTCOMES:
Change in total score of self-reported daytime sleepiness using Epworth Sleepiness Scale | 5 weeks
  Sleep satisfaction will be self-recorded on Epworth Sleepiness Scale (ESS). Range from 0 equal to lowest sleepiness during day and 24 equal to highest sleepiness during day.
Change in total score of self-reported sleep quality on Pittsburgh Quality Index | 5 weeks
  Range is from 0-21 with 0 equal to better sleep quality and 21 meaning worst sleep quality.
Change in total score for sleep quality with Post Polysomnogram Sleep Assessment | 5 weeks
  Sleep quality will be recorded from range 5 to 30 total score, 5 equal to worst sleep quality and 30 equal to best sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Jain, MD, Principal Investigator — George Washington University; David Mendelowitz, PhD, Principal Investigator — George Washington University
Locations (1):
- Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No